CLINICAL TRIAL: NCT00105443
Title: A Phase III Randomized, Placebo-controlled Study of Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Phase III Study of Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Acronym: SHARP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100554; 2004-001773-26 (EudraCT Number)
Record Dates: First submitted 2005-03-14; First posted 2005-03-15 (Estimated); Results first posted 2010-09-27 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Liver Cancer; Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Sorafenib 400 mg was administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily; 2 dose reductions to predefined levels of 400 mg once daily (OD) and 400 mg every other day were permitted for adverse events related to study treatment. Follow-up / Open Label phase: Subjects on sorafenib who continued the study, continued on the same dose of sorafenib as during the double-blind study.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Placebo (Placebo Comparator): Sorafenib-matching placebo tablets were orally administered twice daily (bid). Follow-up / Open Label phase: Subjects on placebo who chose to switch to sorafenib, received an oral dose of 400 mg (2 x 200 mg tablets) bid; similar to the double-blind study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib 400 mg was administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid); 2 dose reductions to predefined levels of 400 mg once daily (OD) and 400 mg every other day were permitted for adverse events related to study treatment.
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Placebo — Sorafenib-matching placebo tablets were orally administered twice daily (bid).
  Arms: Placebo

SUMMARY:
The purpose of the study is: Find out if patients receiving sorafenib will live longer. Find out if sorafenib has any effect on patient reported outcomes. Find out if sorafenib prevents the growth of or shrinks liver tumors and/or their metastases. Determine the pharmacokinetics (PK) in patients with liver cancer.

DETAILED DESCRIPTION:
The following abbreviations were used in the Adverse Event section:

* international normalized ratio (inr)
* Common Terminology Criteria for Adverse Events (ctcae)
* Not Otherwise Specified (nos)
* Gastrointestinal (gi)
* Central nervous system (cns)
* Absolute Neutrophil Count (anc)
* Alanine aminotransferase (ALT)
* Aspartate aminotransferase (AST)
* Creatine phosphokinase (cpk)
* Gammaglutamyltransferase (ggt)
* Genitourinary (gu)
* Atrioventricular (av)

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 18 years and above, Genders eligible for study: both
* Patients who have a life expectancy of at least 12 weeks
* Patients with histologically or cytologically documented Hepatocellular Carcinoma (HCC)
* Patients must have at least one tumor lesion that meets both of the following criteria: (1) Accurately measured in at least one dimension according to RECIST (Response Evaluation Criteria in Solid Tumors) (2) Not previously treated with local therapy
* Patients who have an ECOG (Eastern Cooperative Oncology Group) PS (Performance Status) of 0, 1, or 2

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta [Noninvasive papillary carcinoma], Tis [Carcinoma in situ: "flat tumor"] & T1 [Tumor invades subepithelial connective tissue]). Any cancer curatively treated > 3 years prior to entry is permitted
* Renal failure requiring hemo- or peritoneal dialysis
* History of cardiac disease
* Active clinically serious infections
* Known history of human immunodeficiency virus (HIV) infection
* Known central nervous system tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2005-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (142):
- United States (27):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Los Angeles, California
  - Orange, California
  - San Francisco, California
  - Stanford, California
  - Farmington, Connecticut
  - New Haven, Connecticut
  - Gainesville, Florida
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Manhasset, New York
  - New York, New York
  - Canton, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Richmond, Virginia
  - Seattle, Washington
- Argentina (5):
  - Mar del Plata, Buenos Aires
  - Pilar, Buenos Aires
  - Bueno Aires, Ciudad Auton. de Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - San Miguel de Tucumán, Tucumán Province
- Australia (6):
  - Camperdown, New South Wales
  - Randwick, New South Wales
  - Westmead, New South Wales
  - East Bentleigh, Victoria
  - Heidelberg, Victoria
  - Melbourne, Victoria
- Belgium (4):
  - Bruges
  - Bruxelles - Brussel
  - Ghent
  - Leuven
- Brazil (3):
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Belo Horizonte
- Bulgaria (3):
  - Sofia
  - Stara Zagora
  - Varna
- Canada (8):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Chile (3):
  - Santiago, Santiago Metropolitan
  - Santiago
  - Santiago Región Metropolitana
- Zagreb, Croatia
- France (10):
  - Bondy
  - Bordeaux
  - Clichy
  - Dijon
  - Lille
  - Marseille
  - Nantes
  - Paris
  - Rennes
  - Vandœuvre-lès-Nancy
- Germany (15):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Hanover, Lower Saxony
  - Bonn, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
- Greece (5):
  - Haidari, Attica
  - Thessaloniki, Thessaloniki
  - Athens
  - Ioannina
  - Thessaloniki
- Israel (4):
  - Petah Tikva, Israel
  - Tel Aviv, Israel
  - Zrifin, Israel
  - Haifa
- Italy (10):
  - Forlì, Forlì
  - Rozzano, Milano
  - Avellino
  - Bologna
  - Milan
  - Padua
  - Palermo
  - Pavia
  - Pisa
  - Roma
- Mexico (3):
  - Mexico City, Mexico City
  - México, D.F.
  - Monterrey
- New Zealand (2):
  - Auckland
  - Wellington South
- Peru (3):
  - Comas Lima
  - Lima
  - Lima Cercado
- Poland (3):
  - Gdansk
  - Poznan
  - Warsaw
- Romania (3):
  - Iași, Iaşi
  - Timișoara, Timiș County
  - Craiova Dolj
- Russia (7):
  - Kazan'
  - Kirov
  - Krasnodar
  - Moscow
  - Saint Petersburg
  - Tolgliatti
  - Yekaterinburg
- Spain (8):
  - Alicante, Alicante
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Cruces/Barakaldo, Bilbao
  - Córdoba, Córdoba
  - Madrid, Madrid
  - Pamplona, Pamplona
  - Valencia, Valencia
- Switzerland (4):
  - Bern, Canton of Bern
  - Geneva, Canton of Geneva
  - Sankt Gallen, Canton of St. Gallen
  - Zurich, Canton of Zurich
- United Kingdom (5):
  - Bristol, Avon
  - London, London
  - Oxford, Oxfordshire
  - Glasgow, Stratchclyde
  - Newcastle upon Tyne

REFERENCES:
- [Result] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Derived] Wu W, Mao H, Song J, Yang F. Bibliometric analysis of hepatocellular carcinoma and tyrosine kinase inhibitors. Medicine (Baltimore). 2025 May 16;104(20):e42015. doi: 10.1097/MD.0000000000042015. PMID 40388796
- [Derived] Bruix J, Cheng AL, Meinhardt G, Nakajima K, De Sanctis Y, Llovet J. Prognostic factors and predictors of sorafenib benefit in patients with hepatocellular carcinoma: Analysis of two phase III studies. J Hepatol. 2017 Nov;67(5):999-1008. doi: 10.1016/j.jhep.2017.06.026. Epub 2017 Jul 4. PMID 28687477
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with advanced hepatocellular carcinoma (HCC) were enrolled from Mar 10, 2005 to Apr 11, 2006 at 121 study centers in 21 countries around the Globe.
Pre-assignment Details: After a 28 day screening period (902 subjects), 602 were randomized to Sorafenib (400 mg) twice daily (bid), or matching placebo. Majority of screen failures did not meet inclusion criteria. Efficacy population (intent-to-treat, ITT) was all randomized subjects (602), safety population was all subjects receiving at least 1 dose of study drug (599).
Groups:
- A1) Sorafenib (Nexavar, BAY43-9006) - no Open Label Phase: Sorafenib 400 mg was administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily; 2 dose reductions to predefined levels of 400 mg once daily (OD) and 400 mg every other day were permitted for adverse events related to study treatment. Note: Safety Data of participants in the arm presented here are reported in Reporting Groups (RG) RG1 and RG3 in the Safety section.
- A2) Sorafenib (Nexavar, BAY43-9006) - With Open Label Phase: Sorafenib 400 mg was administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily; 2 dose reductions to predefined levels of 400 mg once daily (OD) and 400 mg every other day were permitted for adverse events related to study treatment. Follow-up / Open Label phase: Subjects on sorafenib who continued the study, continued on the same dose of sorafenib as during the double-blind study Note: Safety Data of participants in the arm presented here are reported in Reporting Groups (RG) RG1 and RG3 in the Safety section.
- B1) Placebo - no Open Label Phase: Sorafenib-matching placebo tablets were orally administered twice daily (bid).
  Note: Safety Data of participants in the arm presented here are reported in Reporting Groups (RG) RG2 and RG4 in the Safety section.
- B2) Placebo First - Then Open Label Sorafenib Treatment Phase: Sorafenib-matching placebo tablets were orally administered twice daily (bid). Follow-up / Open Label phase: Subjects on placebo who chose to switch to sorafenib, received an oral dose of 400 mg (2 x 200 mg tablets) bid; similar to the double-blind study.
  Note: Safety Data of participants in the arm presented here are reported in Reporting Groups (RG) RG2, RG4, and RG5 in the Safety section.
Period: Double-Blind Treatment
Arm/Group | A1) Sorafenib (Nexavar, BAY43-9006) - no Open Label Phase | A2) Sorafenib (Nexavar, BAY43-9006) - With Open Label Phase | B1) Placebo - no Open Label Phase | B2) Placebo First - Then Open Label Sorafenib Treatment Phase
Started | 242 | 57 | 256 | 47
Received Treatment | 240 (Subjects at Risk/Safety Population - partly in RG1 and RG3 (RG = Reporting Group for Safety Data)) | 57 (Subjects at Risk/Safety Population - partly in RG1 and RG3) | 255 (Subjects at Risk/Safety Population - partly in RG2 and RG4) | 47 (Subjects at Risk/Safety Population - partly in RG2 and RG4 as well as RG5)
Completed | 228 (228 participants directly switched to the Follow-up (FU) phase only) | 57 (47 participants continued with Sorafenib Open Label (OL); 10 first to FU prior to also switch to OL) | 245 (245 participants directly switched to the Follow-up (FU) phase) | 47 (36 participants switched to Sorafenib Open Label (OL); 11 first to FU prior to also switch to OL)
Not Completed | 14 | 0 | 11 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 7 | 0
Not completed — Physician Decision | 1 | 0 | 2 | 0
Not completed — Radiological and symptomatic progression | 4 | 0 | 1 | 0
Period: Follow-up and/or Open Label Nexavar
Arm/Group | A1) Sorafenib (Nexavar, BAY43-9006) - no Open Label Phase | A2) Sorafenib (Nexavar, BAY43-9006) - With Open Label Phase | B1) Placebo - no Open Label Phase | B2) Placebo First - Then Open Label Sorafenib Treatment Phase
Started | 228 (At start of period, 228 participants directly switched to Follow-up (FU)) | 57 (At start of period, 47 participants directly switched to Open Label (OL) Sorafenib treatment) | 245 (At start of period, 245 participants directly switched to Follow-up (FU)) | 47 (At start of period, 36 participants directly switched to Open Label (OL) Sorafenib treatment)
Follow-up Only (no Open Label Treatment) | 228 (In parallel to "Open Label treatment only" phase) | 0 | 245 (In parallel to "Open Label treatment only" phase) | 0
Open Label Treatment Only (no Follow-up) | 0 | 47 (In parallel to "Follow-up only" phase; participants received Sorafenib 400 mg bid) | 0 | 36 (In parallel to "Follow-up only" phase; participants received Sorafenib 400 mg bid)
Follow-up First, Then Open Label | 0 | 10 | 0 | 11
Completed | 0 | 0 (57 participants in total (47 + 10) received Open Label Sorafenib treatment (Subjects at Risk)) | 0 | 0 (47 participants in total (36 + 11) received Open Label Sorafenib treatment (Subjects at Risk))
Not Completed | 228 | 57 | 245 | 47
Not completed — Death | 180 | 7 | 219 | 4
Not completed — Lost to Follow-up | 14 | 0 | 10 | 0
Not completed — Withdrawal by Subject | 24 | 3 | 13 | 4
Not completed — Adverse Event | 0 | 14 | 0 | 16
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0
Not completed — Progression by clinical judgment | 0 | 2 | 0 | 5
Not completed — Progression, measurement proven | 0 | 3 | 0 | 3
Not completed — Disease progression, recurrence, relapse | 6 | 0 | 1 | 0
Not completed — Endpoint record not completed | 2 | 2 | 1 | 2
Not completed — Planned switch to OL; record incomplete | 1 | 0 | 0 | 0
Not completed — Non-compliant with study medication | 0 | 0 | 0 | 1
Not completed — Reached ECOG 4 | 0 | 1 | 0 | 1
Not completed — Switch to commercial drug | 0 | 23 | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Total
Number analyzed (Participants) | 299 | 303 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (11.2) | 66.3 (10.2) | 65.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 260 | 264 | 524
Baseline Eastern Cooperative Oncology Group (ECOG) [Number; unit: participants] — Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is a scale that measures how cancer affects a patient. The scale ranges from 0 (fully active) to 5 (dead). Subjects entering this study were to have an ECOG score of 0, 1 or 2.
  participants
    0 = fully active | 161 | 164 | 325
    1 = restricted in physical activity but ambulatory | 114 | 117 | 231
    2 = capable of selfcare | 24 | 22 | 46
Tumor burden [Number; unit: participants] — Tumor burden refers to the number of cancer cells, the size of a tumor, or the amount of cancer in the body and is also called the tumor load. Randomization was stratified by "tumor burden" assessment, ie, the presence of either macroscopic vascular invasion as determined by radiological assessment and/or extra-hepatic spread versus none.
  participants
    Absent | 90 | 91 | 181
    Present | 209 | 212 | 421

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from date of starting treatment to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Time Frame: from randomization to death due to any cause until an average 7.2 months later up to the data cut-off date approximately 19 months after start of enrollment
Population: In this study the overall survival was measured for the ITT population from the date of randomization until the date of death due to any cause. For patients alive or lost to follow-up at the time of analysis, time to death was to be censored at their last date of follow-up, or at the data cut-off of 17 Oct 2006.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 299 | 303
days | 324 [286 to 405] | 241 [206 to 276]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; The 2 arms were compared using a 1-sided log-rank test with an overall alpha of 0.02 stratified by region, ECOG PS and "tumor burden". In addition to the final analysis at the end of the study, 2 formal interim analyses of overall survival were planned. An alpha spending function was used to ensure that the false positive rate is less than or equal to 0.02 (1-sided). The study was stopped at the second interim analysis, the results of which are reported here; Test type: Superiority or Other; p = 0.00583, Log Rank — According to the pre-specified O'Brien-Fleming alpha spending function, the alpha value for this second interim analysis was 0.0073 (corresponding to a nominal value of 0.0077 after taking into account the first interim analysis); Hazard Ratio (HR) = 0.6931, 95% CI [0.5549 to 0.8658] — This is the sorafenib to placebo hazard ratio

2. Primary Outcome: Time to Symptomatic Progression (TTSP)
Description: TTSP was defined as the time from randomization to the first documented symptomatic progression.
Time Frame: from randomization to the first documented symptomatic progression until an average 4.8 months later up to the data cut-off date approximately 19 months after start of enrollment
Population: This analysis was for the ITT population. For subjects who had not progressed symptomatically at the time of interim analysis, TTSP was censored at the date of their last Functional Assessment of Cancer Therapy (FACT) Hepatobiliary Symptom Index (FHSI-8) questionnaire assessment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 299 | 303
days | 126 [105 to 126] | 148 [129 to 192]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; The 2 arms were compared using a 1-sided log-rank test with an overall alpha of 0.005 stratified by region, ECOG PS and "tumor burden". This was a co-primary endpoint with overall survival. No alpha-spending adjustments were necessary as it was only to be analyzed at the end of study; Test type: Superiority or Other; p = 0.7676, Log Rank; Hazard Ratio (HR) = 1.0764, 95% CI [0.8837 to 1.3110] — This is the sorafenib to placebo hazard ratio

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from randomization to disease progression (radiological only). Subjects without tumor progression at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: from randomization to disease progression based on radiological assessment until an average 2.8 months later up to the data cut-off date approximately 19 months after start of enrollment
Population: The primary analysis of TTP for the ITT population was based on the independent radiological review for the interim analysis. The cut-off date chosen for the analysis of radiological progression events was 12 May 2006
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 299 | 303
days | 168 [126 to 210] | 86 [82 to 120]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; In the analysis of TTP, based on independent radiological review performed to review data up to 12 May 2006, the 2 treatment groups were compared using a 1-sided log rank test with an alpha of 0.025, stratified by region, ECOG PS, and "tumor burden"; Test type: Superiority or Other; p = 0.000007, Log Rank; Hazard Ratio (HR) = 0.5764, 95% CI [0.4484 to 0.7410] — This is the sorafenib to placebo hazard ratio

4. Secondary Outcome: Disease Control (DC)
Description: The DC is defined as the number of subjects with a best response rating of complete response (CR), partial response (PR), or stable disease (SD) that is maintained at least 28 days from the first manifestation of that rating. Definitions: CR = disappearance of all clinical and radiological tumor lesions; PR = at least 30% decrease in sum of the longest diameters of tumor lesions; SD = neither sufficient shrinkage to qualify for PR nor sufficient increase for progressive disease.
Time Frame: time from randomization to end of treatment up to the data cutoff date approximately 19 months after start of enrollment
Population: In this study, the DC for the ITT population was determined by independent radiological review and also by investigator assessment (both by using response evaluation criteria in solid tumors [RECIST])
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 299 | 303
Participants | 130 | 96
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Disease control rates were compared between treatment groups using the Cochran Mantel Haenszel (CMH) test with a 1-sided alpha of 0.025, adjusting for region, ECOG PS, and "tumor burden"; Test type: Superiority or Other; p = 0.001641, Cochran-Mantel-Haenszel; Risk Difference (RD) = -11.95, 95% CI [-19.56 to -4.35] — Sorafenib minus placebo difference

5. Secondary Outcome: Patients Reported Outcome (PRO) by Use of the FACT-Hep Questionnaire
Description: PRO is a disease-specific measure, developed as symptom-focused approach in HCC and measured by the response rates for the PWB and FWB subscales of the 45-item Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaire. The FACT-Hep response rate was based on the number of subjects who achieved the 8-point minimally important difference (MID) for this subscale. FACT-Hep total score ranges from 0 to 180, where the highest score represents a maximum achievable quality of life (QoL) value.
Time Frame: from randomization to end of treatment up to the data cutoff date approximately 19 months after start of enrollment
Population: In this study, the PRO was a tertiary efficacy variable assessed for the ITT population at Cycle 3 day 1 or, for those discontinuing prior to that visit, at end of study. It was summarized as number of patients with change from baseline <8 or ≥8 points for each treatment group up to the cutoff date of 17 Oct 2006
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 174 | 178
Participants
  Cycle 3 day 1 change <8 points | 151 | 139
  Cycle 3 day 1 change ≥8 points | 23 | 39

6. Post Hoc Outcome: Overall Survival
Description: as for outcome 1
Time Frame: from randomization to death due to any cause until an average 8.5 months later up to the data cut-off date approximately 23 months after start of enrollment
Population: The OS data (ITT population) are descriptive only (no p-values) from the date of randomization to the date of death due to any cause. For patients alive at the time of analysis, time to death was censored at the date of last follow-up or at the data cutoff date of 09 Feb 2007 when subjects were given the option to crossover to sorafenib treatment
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 299 | 303
Days | 327 [287 to 400] | 243 [206 to 289]

7. Post Hoc Outcome: Time to Symptomatic Progression (TTSP)
Description: TTSP was defined as the time from randomization to the first documented symptomatic progression
Time Frame: from randomization to the first documented symptomatic progression until an average 5.7 months later up to the data cut-off date approximately 23 months after start of enrollment
Population: For subjects (in the ITT population) who had not progressed symptomatically at the time of interim analysis, TTSP was censored at the date of last FACT FHSI-8 questionnaire assessment (upon an interim review by the Data Monitoring Committee on 09 Feb 2007), when the study was considered positive for its primary endpoint, OS, and was stopped early.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 299 | 303
Days | 127 [106 to 152] | 148 [132 to 195]

8. Post Hoc Outcome: Time to Progression (TTP)
Description: as for outcome 3
Time Frame: from randomization to disease progression based on radiological assessment until an average 2.8 months later up to the data cut-off date approximately 23 months after start of enrollment
Population: The independent radiological review as initially scheduled for the interim analysis did not continue after 12 May 2006. The primary analysis of TTP for the ITT population after 12 May 2006 up to the cutoff date of 09 Feb 2007 was based on the Investigator radiological assessments
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 299 | 303
Days | 168 [126 to 210] | 86 [82 to 120]

9. Post Hoc Outcome: Disease Control (DC)
Description: The DC is defined as the number of subjects with a best response rating of CR, PR, or SD that is maintained at least 28 days from the first manifestation of that rating.
Time Frame: from randomization to end of treatment up to the data cutoff date approximately 23 months after start of enrollment
Population: The disease control rate for the ITT population was determined by independent radiological review and also by investigator assessment (both by using response evaluation criteria in solid tumors (RECIST) up to the cutoff date of 09 Feb 2007
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 299 | 303
Participants | 130 | 96

10. Post Hoc Outcome: Patients Reported Outcome (PRO) by Use of the FACT-Hep Questionnaire
Description: PRO is a disease-specific measure, developed as symptom-focused approach in HCC and measured by the response rates for the PWB and FWB subscales of the 45-item Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaire. The FACT-Hep response rate was based on the number of subjects who achieved the 8-point minimally important difference (MID) for this subscale. FACT-Hep total score ranges from 0 to 180, where the highest score represents a maximum achievable quality of life (QoL) value. At the cut-off date for this analysis, one more patient data has been gained.
Time Frame: from randomization to end of treatment up to the data cutoff date approximately 23 months after start of enrollment
Population: In this study, the PRO was a tertiary efficacy variable assessed for the ITT population at Cycle 3 Day 1 or, for those discontinuing prior to that visit, at the end of study. It was summarized as number of patients with change from baseline <8 to ≥8 points for each treatment group up to the cutoff date of 09 Feb 2007.
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 174 | 179
Participants
  Cycle 3 day 1 change <8 points | 151 | 139
  Cycle 3 day 1 change ≥8 points | 23 | 40

ADVERSE EVENTS:
Time Frame: Reporting Group (RG) 1 + 2: Data for Interim Analysis, cut-off Oct 17, 2006; RG 3: Data during and after unblinding (until Nov 21, 2008); RG 4: Data prior to date of unblinding (Feb 9, 2007); RG 5: Data after unblinding (Open Label; until Nov 21, 2008)
Description: RG 1 + 3 description: All subjects randomized to Sorafenib treatment; RG 2 + 4 description: All subjects randomized to Placebo before unblinding (when they were on Placebo, before they had the opportunity to switch to Sorafenib treatment); RG 5 description: All placebo subjects who switched to Sorafenib treatment after unblinding occurred.
Groups:
- Sorafenib (Nexavar) Arm Double-Blind Phase (Interim Data Only): Reporting Group 1 (RG 1): All participants in Double-Blind phase randomized to Sorafenib treatment (data before Oct 17, 2006); Sorafenib 400 mg was administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid); 2 dose reductions to predefined levels of 400 mg once daily (OD) and 400 mg every other day were permitted for adverse events related to study treatment. Note: Safety Data presented here include participants listed in Arms A1 and A2 of the Participant Flow section.
- Placebo Arm Double-Blind Phase (Interim Data Only): Reporting Group 2 (RG 2): All participants in Double-Blind phase randomized to Sorafenib-matching placebo (data before Oct 17, 2006); Sorafenib-matching placebo tablets were orally administered twice daily (bid).
  Note: Safety Data presented here include participants listed in Arms B1 and B2 of the Participant Flow section.
- Sorafenib (Nexavar) Arm Complete (Incl. Open Label Phase): Reporting Group 3 (RG 3): All participants that initially were randomized to Sorafenib treatment (data before unblinding (= Double-Blind phase) and after unblinding (= Open Label phase)), until Nov 21, 2008); Sorafenib 400 mg was administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid); 2 dose reductions to predefined levels of 400 mg once daily (OD) and 400 mg every other day were permitted for adverse events related to study treatment. Note: Safety Data presented here include participants listed in Arms A1 and A2 of the Participant Flow section.
- Placebo Arm, Complete Double-Blind Phase: Reporting Group 4 (RG 4): All participants that initially were randomized to Placebo (data from Placebo patients before unblinding at Feb 09, 2007); Sorafenib-matching placebo tablets were orally administered twice daily (bid).
  Note: Safety Data presented here include participants listed in Arms B1 and B2 of the Participant Flow section.
- Subjects Switching From Placebo to Sorafenib (Open Label Only): Reporting Group 5 (RG 5): Participants initially randomized to Placebo who switched to Sorafenib in Open Label phase (data after unblinding only, from Feb 09, 2007 until Nov 21, 2008); Sorafenib 400 mg was administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid). Note: Safety Data presented here include participants listed in Arm B2 of the Participant Flow section.
Arm/Group | Sorafenib (Nexavar) Arm Double-Blind Phase (Interim Data Only) | Placebo Arm Double-Blind Phase (Interim Data Only) | Sorafenib (Nexavar) Arm Complete (Incl. Open Label Phase) | Placebo Arm, Complete Double-Blind Phase | Subjects Switching From Placebo to Sorafenib (Open Label Only)
Serious Adverse Events (participants affected / at risk) | 153/297 | 164/302 | 191/297 | 185/302 | 26/47
Other Adverse Events (participants affected / at risk) | 275/297 | 259/302 | 281/297 | 271/302 | 43/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar) Arm Double-Blind Phase (Interim Data Only) (N=297) | Placebo Arm Double-Blind Phase (Interim Data Only) (N=302) | Sorafenib (Nexavar) Arm Complete (Incl. Open Label Phase) (N=297) | Placebo Arm, Complete Double-Blind Phase (N=302) | Subjects Switching From Placebo to Sorafenib (Open Label Only) (N=47)
neutrophils (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
hemoglobin (Blood and lymphatic system disorders) | 8 | 6 | 11 | 7 | 0
leukocytes (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
supraventricular arrhythmia, atrial fibrillation (Cardiac disorders) | 1 | 2 | 1 | 3 | 0
conduction abnormality, av block - first degree (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
supraventricular arrhythmia, sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
ventricular arrhythmia, ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
ventricular arrhythmia, ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
inr (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0
left ventricular diastolic dysfunction (Cardiac disorders) | 2 | 0 | 2 | 0 | 0
hypertension (Cardiac disorders) | 1 | 1 | 1 | 1 | 0
cardiac ischemia/infarction (Cardiac disorders) | 8 | 4 | 9 | 5 | 1
hypotension (Cardiac disorders) | 1 | 2 | 1 | 1 | 0
cardiac general - other (Cardiac disorders) | 0 | 3 | 0 | 3 | 0
right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
left ventricular systolic dysfunction (Cardiac disorders) | 1 | 2 | 2 | 2 | 0
death not associated with ctcae term, death nos (General disorders) | 1 | 4 | 1 | 5 | 1
death not associated with ctcae term, disease progression nos (General disorders) | 56 | 61 | 68 | 66 | 10
death not associated with ctcae term, multi-organ failure (General disorders) | 1 | 0 | 4 | 0 | 0
death not associated with ctcae term, sudden death (General disorders) | 0 | 1 | 1 | 1 | 1
hyperthyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0
fever (General disorders) | 3 | 4 | 4 | 4 | 1
insomnia (General disorders) | 0 | 1 | 0 | 0 | 0
fatigue (General disorders) | 5 | 9 | 7 | 6 | 1
weight loss (General disorders) | 0 | 3 | 0 | 1 | 0
constitutional symptoms - other (General disorders) | 3 | 6 | 6 | 8 | 2
anorexia (Gastrointestinal disorders) | 3 | 1 | 3 | 1 | 0
ascites (Gastrointestinal disorders) | 14 | 13 | 16 | 20 | 4
colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
dehydration (Gastrointestinal disorders) | 9 | 1 | 10 | 1 | 0
diarrhea (Gastrointestinal disorders) | 14 | 5 | 16 | 5 | 1
dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
nausea (Gastrointestinal disorders) | 0 | 4 | 0 | 3 | 0
gi - other (Gastrointestinal disorders) | 4 | 0 | 6 | 0 | 1
perforation, gi, colon (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
stricture, gi, biliary tree (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
ulcer, gi, duodenum (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
ulcer, gi, stomach (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
vomiting (Gastrointestinal disorders) | 5 | 4 | 5 | 4 | 0
cns hemorrhage (Vascular disorders) | 2 | 1 | 2 | 1 | 0
hematoma (Vascular disorders) | 0 | 1 | 0 | 1 | 0
hemorrhage, gi, abdomen nos (Vascular disorders) | 2 | 3 | 2 | 3 | 0
hemorrhage, gi, colon (Vascular disorders) | 1 | 0 | 1 | 0 | 0
hemorrhage, gi, duodenum (Vascular disorders) | 1 | 2 | 1 | 3 | 0
hemorrhage, gi, esophagus (Vascular disorders) | 2 | 3 | 4 | 4 | 1
hemorrhage, gi, varices (esophageal) (Vascular disorders) | 7 | 11 | 8 | 13 | 1
hemorrhage, gi, stomach (Vascular disorders) | 4 | 2 | 5 | 2 | 0
hemorrhage, gi, liver (Vascular disorders) | 4 | 1 | 6 | 1 | 0
hemorrhage, gi, lower gi nos (Vascular disorders) | 0 | 1 | 0 | 1 | 0
hemorrhage, gi, oral cavity (Vascular disorders) | 0 | 1 | 0 | 1 | 0
hemorrhage, gi, peritoneal cavity (Vascular disorders) | 0 | 6 | 2 | 8 | 0
hemorrhage, gi, varices (rectal) (Vascular disorders) | 1 | 0 | 1 | 0 | 0
hemorrhage, gi, upper gi nos (Vascular disorders) | 3 | 6 | 5 | 6 | 0
hemorrhage with surgery (Vascular disorders) | 0 | 1 | 0 | 1 | 0
hemorrhage - other (Vascular disorders) | 1 | 1 | 2 | 1 | 0
hemorrhage pulmonary, lung (Vascular disorders) | 1 | 0 | 1 | 0 | 0
hemorrhage pulmonary, pleura (Vascular disorders) | 0 | 1 | 0 | 1 | 0
cholecystitis (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0
liver dysfunction (Gastrointestinal disorders) | 21 | 14 | 21 | 18 | 1
hepatobiliary - other (Gastrointestinal disorders) | 11 | 16 | 16 | 22 | 5
pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
infection (documented clinically), abdomen nos (Infections and infestations) | 1 | 0 | 1 | 0 | 0
infection (documented clinically), anal/perianal (Infections and infestations) | 1 | 0 | 1 | 0 | 0
infection (documented clinically), biliary tree (Infections and infestations) | 0 | 1 | 0 | 1 | 0
infection (documented clinically), lung (pneumonia) (Infections and infestations) | 3 | 3 | 6 | 4 | 2
infection (documented clinically), skin (cellulitis) (Infections and infestations) | 1 | 1 | 1 | 1 | 0
infection (documented clinically), soft tissue nos (Infections and infestations) | 0 | 1 | 0 | 1 | 0
infection (documented clinically), upper airway nos (Infections and infestations) | 1 | 0 | 1 | 0 | 0
infection (documented clinically), urinary tract nos (Infections and infestations) | 3 | 0 | 3 | 0 | 0
infection with normal anc, bronchus (Infections and infestations) | 0 | 1 | 0 | 1 | 0
infection with normal anc, gallbladder (cholecystitis) (Infections and infestations) | 1 | 0 | 1 | 0 | 0
infection with normal anc, oral cavity-gums (gingivitis) (Infections and infestations) | 0 | 1 | 0 | 1 | 0
infection with normal anc, peritoneal cavity (Infections and infestations) | 0 | 2 | 0 | 2 | 0
infection with normal anc, skin (cellulitis) (Infections and infestations) | 0 | 1 | 0 | 1 | 0
infection with normal anc, urinary tract nos (Infections and infestations) | 0 | 1 | 0 | 1 | 0
infection - other (Infections and infestations) | 0 | 3 | 2 | 4 | 0
infection with unknown anc, biliary tree (Infections and infestations) | 1 | 0 | 1 | 0 | 0
infection with unknown anc, lung (pneumonia) (Infections and infestations) | 0 | 3 | 0 | 4 | 0
infection with unknown anc, peritoneal cavity (Infections and infestations) | 1 | 2 | 1 | 2 | 0
infection with unknown anc, urinary tract nos (Infections and infestations) | 0 | 1 | 0 | 1 | 0
infection with unknown anc, wound (Infections and infestations) | 1 | 0 | 1 | 0 | 0
edema: limb (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0 | 0
lymphatics - other (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
fracture (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5 | 4 | 1
musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 3 | 0
device/prosthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
muscle weakness, whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
ALT (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0
AST (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 0
cpk (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
creatinine (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1
ggt (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 6 | 4 | 6 | 5 | 1
hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 0
hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 0
hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0
hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
hypoglycemia (Metabolism and nutrition disorders) | 5 | 3 | 5 | 3 | 1
hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
cns ischemia (Nervous system disorders) | 0 | 4 | 1 | 4 | 2
confusion (Nervous system disorders) | 1 | 1 | 1 | 1 | 0
dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
encephalopathy (Nervous system disorders) | 2 | 2 | 4 | 3 | 1
mood alteration, depression (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
neuropathy: motor (Nervous system disorders) | 1 | 3 | 1 | 3 | 0
neurology - other (Nervous system disorders) | 0 | 3 | 0 | 3 | 0
neuropathy: sensory (Nervous system disorders) | 1 | 1 | 1 | 1 | 0
seizure (Nervous system disorders) | 1 | 2 | 1 | 2 | 0
somnolence (Nervous system disorders) | 2 | 2 | 2 | 2 | 0
syncope (fainting) (Nervous system disorders) | 2 | 0 | 2 | 0 | 0
retinal detachment (Eye disorders) | 0 | 1 | 0 | 1 | 0
pain, back (General disorders) | 3 | 3 | 3 | 4 | 0
pain, extremity-limb (General disorders) | 1 | 0 | 1 | 0 | 0
pain, tumor pain (General disorders) | 1 | 1 | 2 | 1 | 0
pain, abdomen nos (General disorders) | 7 | 8 | 10 | 9 | 0
pain, joint (General disorders) | 3 | 0 | 3 | 1 | 0
pain, bone (General disorders) | 3 | 1 | 3 | 1 | 0
pain, other (General disorders) | 1 | 0 | 1 | 0 | 0
pain, liver (General disorders) | 0 | 2 | 0 | 3 | 0
pain, neuralgia/peripheral nerve (General disorders) | 0 | 1 | 0 | 1 | 0
pain, stomach (General disorders) | 0 | 1 | 0 | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 1
hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 2 | 0
renal failure (Renal and urinary disorders) | 1 | 8 | 2 | 8 | 1
obstruction, gu, ureter (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0
dermatology - other (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
intraop injury, biliary tree - common bile duct (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
syndromes - other (General disorders) | 2 | 0 | 1 | 0 | 0
peripheral arterial ischemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0
thrombosis/thrombus/embolism (Vascular disorders) | 3 | 3 | 7 | 5 | 1
visceral arterial ischemia (Vascular disorders) | 1 | 1 | 1 | 1 | 0
not coded yet (General disorders) | 0 | 1 | 0 | 0 | 0
conduction abnormality, asystole (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
conduction abnormality, av block-3rd degree (complete av block (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
cardiac arrhythmia - other (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
cardiopulmonary arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
obstruction, gi, small bowel nos (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
perforation, gi, appendix (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
hemorrhage, gi, rectum (Vascular disorders) | 0 | 0 | 1 | 0 | 1
infection (documented clinically), blood (Infections and infestations) | 0 | 0 | 1 | 0 | 0
infection with normal anc, anal/perianal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
infection with normal anc, appendix (Infections and infestations) | 0 | 0 | 1 | 0 | 0
infection with normal anc, pancreas (Infections and infestations) | 0 | 0 | 1 | 0 | 0
infection with unknown anc, appendix (Infections and infestations) | 0 | 0 | 1 | 0 | 0
infection with unknown anc, blood (Infections and infestations) | 0 | 0 | 0 | 0 | 1
infection with unknown anc, bronchus (Infections and infestations) | 0 | 0 | 1 | 0 | 0
lymphedema-related fibrosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
edema: head and neck (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
cognitive disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
pain, chest/thorax nos (General disorders) | 0 | 0 | 0 | 1 | 0
urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
decubitus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
tumor flare (General disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar) Arm Double-Blind Phase (Interim Data Only) (N=297) | Placebo Arm Double-Blind Phase (Interim Data Only) (N=302) | Sorafenib (Nexavar) Arm Complete (Incl. Open Label Phase) (N=297) | Placebo Arm, Complete Double-Blind Phase (N=302) | Subjects Switching From Placebo to Sorafenib (Open Label Only) (N=47)
hemoglobin (Blood and lymphatic system disorders) | 25 | 22 | 36 | 25 | 5
hypertension (Cardiac disorders) | 27 | 12 | 32 | 13 | 6
fever (General disorders) | 29 | 28 | 35 | 30 | 2
insomnia (General disorders) | 21 | 22 | 26 | 23 | 5
fatigue (General disorders) | 133 | 132 | 145 | 144 | 23
weight loss (General disorders) | 89 | 28 | 93 | 31 | 10
anorexia (Gastrointestinal disorders) | 83 | 52 | 89 | 56 | 8
ascites (Gastrointestinal disorders) | 61 | 67 | 80 | 67 | 9
constipation (Gastrointestinal disorders) | 41 | 31 | 44 | 32 | 3
diarrhea (Gastrointestinal disorders) | 158 | 74 | 166 | 82 | 22
heartburn (Gastrointestinal disorders) | 15 | 10 | 16 | 10 | 1
mucositis (functional/symptomatic), oral cavity (Gastrointestinal disorders) | 15 | 6 | 16 | 8 | 0
mucositis (clinical exam), oral cavity (Gastrointestinal disorders) | 16 | 10 | 19 | 10 | 1
nausea (Gastrointestinal disorders) | 71 | 58 | 73 | 63 | 8
gi - other (Gastrointestinal disorders) | 16 | 10 | 22 | 13 | 3
vomiting (Gastrointestinal disorders) | 41 | 30 | 48 | 34 | 4
liver dysfunction (Gastrointestinal disorders) | 18 | 9 | 21 | 10 | 1
edema: limb (Blood and lymphatic system disorders) | 45 | 53 | 59 | 57 | 9
musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 24 | 15 | 31 | 18 | 1
AST (Metabolism and nutrition disorders) | 8 | 18 | 9 | 20 | 1
bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 24 | 23 | 28 | 26 | 1
pain, back (General disorders) | 36 | 38 | 47 | 42 | 4
pain, abdomen nos (General disorders) | 91 | 74 | 99 | 80 | 11
pain, head/headache (General disorders) | 26 | 25 | 29 | 25 | 1
pain, joint (General disorders) | 20 | 26 | 20 | 27 | 1
pain, stomach (General disorders) | 21 | 20 | 23 | 21 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 24 | 16 | 26 | 18 | 3
dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 26 | 22 | 33 | 24 | 3
voice changes (Respiratory, thoracic and mediastinal disorders) | 27 | 4 | 27 | 5 | 1
alopecia (Skin and subcutaneous tissue disorders) | 42 | 5 | 46 | 6 | 6
dry skin (Skin and subcutaneous tissue disorders) | 31 | 18 | 31 | 18 | 3
hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 63 | 9 | 67 | 9 | 6
dermatology - other (Skin and subcutaneous tissue disorders) | 26 | 12 | 30 | 15 | 5
pruritus (Skin and subcutaneous tissue disorders) | 40 | 33 | 44 | 35 | 5
rash/desquamation (Skin and subcutaneous tissue disorders) | 55 | 42 | 59 | 46 | 6
platelets (Blood and lymphatic system disorders) | 9 | 7 | 15 | 8 | 0
constitutional symptoms - other (General disorders) | 7 | 10 | 12 | 12 | 4
dry mouth (Gastrointestinal disorders) | 12 | 9 | 14 | 9 | 3
hemorrhoids (Gastrointestinal disorders) | 7 | 2 | 8 | 3 | 3
hepatobiliary - other (Gastrointestinal disorders) | 12 | 14 | 17 | 17 | 2
infection - other (Infections and infestations) | 6 | 3 | 16 | 6 | 8
mood alteration, depression (Nervous system disorders) | 10 | 7 | 14 | 9 | 7
pain, bone (General disorders) | 12 | 13 | 16 | 15 | 0
pain, liver (General disorders) | 12 | 13 | 13 | 16 | 1
erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 4 | 3
flu-like syndrome (General disorders) | 8 | 7 | 9 | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less